CLINICAL TRIAL: NCT05106803
Title: Antibiotic Profile of Pathogenic Bacteria Isolated From Postsurgical Site Infections in Public Hospitals in Northern Jordan
Brief Title: Antibiotic Profile of Pathogenic Bacteria Isolated in Public Hospitals in Northern Jordan
Status: Completed | Type: Observational
Sponsor: Yarmouk University (Other)
Responsible Party: Principal Investigator, Raed M Ennab, Assistant Professor, Yarmouk University
Other Study IDs: Antibiotic profile in Jordan
Record Dates: First submitted 2021-10-24; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Bacterial Infections; Antibiotic Resistant Infection; Surgical Site Infection
Keywords: antimicrobial; hospital; post-surgical infection; surgery
MeSH Terms: conditions — Bacterial Infections; Surgical Wound Infection | interventions — Ciprofloxacin; Trimethoprim, Sulfamethoxazole Drug Combination; Norfloxacin; Erythromycin; Chloramphenicol; Gentamicins; Tetracycline; Vancomycin; Amoxicillin-Potassium Clavulanate Combination; Cefepime; Penicillins; Ampicillin; Clindamycin; Oxacillin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Wound infection: Patients with surgical site infection as diagnosed by the attending physician
  Interventions: Drug: ciprofloxacin

INTERVENTIONS:
Drug: ciprofloxacin — Antibiotics used in vitro n the study
  Other Names: trimethoprim-sulfamethoxazole; norfloxacin; erythromycin; chloramphenicol; gentamicin; tetracycline; vancomycin; amoxicillin/clavulanic acid; cefepime; penicillin; ampicillin; clindamycin; oxacillin

SUMMARY:
The main aim of the study was to identify the various pathogens associated with surgical site infections and their antibiotic susceptibility in a governmental hospital in northern Jordan.

DETAILED DESCRIPTION:
Background: Surgical site infections are hospital-acquired, vary from one hospital to another, and can cause significant postoperative morbidity, mortality, and prolonged hospital stay.

Aim: The main aim of the study was to identify the various pathogens associated with surgical site infections and their antibiotic susceptibility in a governmental hospital in northern Jordan.

Methods: Postsurgical wound samples were collected and processed in a microbiology laboratory using standard microbiological techniques. Antibiotic susceptibility tests were performed using 13 antibiotics covering the gram-positive and gram-negative bacteria using the disc diffusion test.

ELIGIBILITY:
Inclusion Criteria:

* Post-Surgical Wound Infection

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A hospital-based prospective study was carried out in Public-Teaching Hospital in northern Jordan with a total capacity of 400 beds, All patients meet the criteria of getting post-operative wound infections in different surgical wards and ICUs.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Positive culture | August 2019 to October 2019
  Positive swab culture from the wound

SECONDARY OUTCOMES:
Gram stain and type of Bacteria | August 2019 to October 2019
  Gram stain and type of Bacteria grown in culture media
Antibiotic Susceptibility | August 2019 to October 2019
  Antibiotic Susceptibility to the isolated organisms

CONTACTS AND LOCATIONS:
Overall Officials: Raed M Ennab, Principal Investigator — Department of Clinical Sciences, Faculty Of Medicine, Yarmouk University
Locations (1):
- Yarmouk University, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No